CLINICAL TRIAL: NCT00983268
Title: Phase I Trial of Chemoradiation With Capecitabine and Vorinostat in Pancreatic Cancer.
Brief Title: Capecitabine, Vorinostat, and Radiation Therapy in Treating Patients With Nonmetastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Emily Chan, MD, PhD, Assistant Professor of Medicine; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0934; P30CA068485 (NIH); VU-VICC-GI-0934; IRB# 090791; NCCN-M02
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Pancreatic Cancer; Periampullary Adenocarcinoma
Keywords: periampullary adenocarcinoma; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Vorinostat; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: capecitabine; Drug: vorinostat; Radiation: Radiotherapy; Procedure: Surgery to remove tumor

INTERVENTIONS:
Drug: capecitabine — 1000 mg taken by mouth on the days of radiation only.
Drug: vorinostat — Vorinostat will be given by mouth on the day of radiation and then Monday-Friday for two weeks after radiation in these 4 possible doses:
  * Vorinostat,at 100 mg
  * Vorinostat,at 200 mg
  * Vorinostat, at 300 mg
  * Vorinostat, at 400 mg
Radiation: Radiotherapy — High-dose hypofractionated radiotherapy consisting of 3000 cGy in 10 fractions, Monday-Friday for 2 weeks.
Procedure: Surgery to remove tumor — Patients will be assessed for resectability within six weeks of the end of chemoradiation, if resectable, surgery will be performed.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells. Giving capecitabine and vorinostat together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vorinostat when given together with capecitabine and radiation therapy in treating patients with nonmetastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of vorinostat when given in combination with capecitabine and high-dose hypofractionated radiotherapy in patients with nonmetastatic pancreatic cancer.

Secondary

* Determine the safety and side effect profile of this regimen in these patients.
* Determine the response rate in patients treated with this regimen.

Correlative

* Compare pre- and post-treatment whole-cell HDAC-activity levels in peripheral blood mononuclear cell samples.
* Assess chromatin structure and DNA damage in surgical tumor tissue samples.
* Assess proliferation and apoptosis by in vivo imaging.

OUTLINE: This is a dose-escalation study of vorinostat.

Patients receive oral capecitabine twice daily and undergo high-dose hypofractionated radiotherapy once daily on days 1-5 and 8-12. Patients also receive oral vorinostat once daily on days 1-5, 8-12, 15-19, and 22-26 in the absence of disease progression or unacceptable toxicity.

Patients are evaluated for surgery within 6 weeks after completion of chemoradiotherapy. Patients with resectable disease proceed to surgery. Patients with unresectable disease may receive oral vorinostat once daily and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for correlative laboratory studies. Patients also undergo diffusion-weighted MRI for analysis of in vivo tumor cellularity.

After completion of study therapy, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed pancreatic or periampullary cancer.
* Patient must be > 18 years of age.
* Patient may be resectable, borderline resectable, or unresectable but locally advanced as determined by radiographic examination and consultation with a surgical oncologist.
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
* Female patients of childbearing potential must be willing to use birth control. The 2 birth control methods can be either 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy, used throughout the study starting with visit 1. The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner) or sponge. Other methods of contraception such as copper intrauterine device or spermicide may be used. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).Female patient of childbearing potential has a negative serum pregnancy test β-hCG within 7 days prior to receiving the first dose of vorinostat.
* Male patients agree to use an adequate method of contraception for the duration of the study.
* Patient has a life expectancy of at least 12 weeks
* Patient must have adequate organ function as indicated by the following laboratory values:
* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL Hemoglobin ≥ 9 g/dL
* Coagulation
* Prothrombin Time or INR ≤1.5x upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) ≤1.2 times the ULN unless the patient is receiving therapeutic anticoagulation.
* K levels - Normal limits
* Mg levels - Normal limits
* Calculated creatinine *clearance ≥20 mL/min
* Serum total bilirubin ≤ 1.5 X ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN
* Alkaline Phosphatase ≤ 2.5 X ULN

  * Creatinine clearance should be calculated per institutional standard.
* Patient must be capable of understanding and complying with the study protocol and able to give informed consent.
* Measurable disease is not an eligibility requirement.

Exclusion Criteria:

* Prior chemotherapy for pancreatic or periampullary cancer.
* Prior radiation to any area within the planned radiation field. All patients with history of prior radiation to any area must be approved by PI.
* Evidence of distant metastases on imaging.
* History of hypersensitivity to fluoropyrimidines or HDACs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vorinostat when given in combination with capecitabine and radiotherapy | Two weeks after completing radiotherapy

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0 | Six weeks after completing chemo-radiation therpay
Tumor response as assessed by RECIST criteria | Six weeks after completing chemo-radiation therpay
Biological effect | Six weeks after completing chemo-radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chan, M.D, Ph.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/